CLINICAL TRIAL: NCT05438732
Title: A Prospective, Multicenter Clinical Study of the Implantable Miniature Telescope, Model SING in Patients with Central Vision Impairment Associated with End-stage Age-related Macular Degeneration (AMD)
Brief Title: Multicenter Clinical Study of the SING-IMT in Patients with Late-stage AMD
Acronym: CONCERTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VisionCare, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDV-SNG-21-001
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy
Keywords: cataract; best-corrected distance visual acuity
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy; Cataract

STUDY DESIGN:
Intervention Model Description: Effectiveness: one-sided asymptotic normal test Safety: one-sided t-test
Masking Description: since the IMT has a unique appearance in the eye, it cannot be masked to the Investigator or to the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SING-IMT Implanted (Experimental): the implanted eye will be the study eye which receives the SING-IMT. Implantation will occur during routine cataract surgery using a proprietary delivery system (loading cartridge and injector), via an approximately 6.5mm incision
  Interventions: Device: smaller incision, new generation implantable miniature telescope (SING-IMT)

INTERVENTIONS:
Device: smaller incision, new generation implantable miniature telescope (SING-IMT) — The IMT (model SING) is an intraocular implant comprised of 2 micro lenses in a glass tube (optics) in a flexible silicone carrier (haptics)

SUMMARY:
The objective of this study is to determine the safety and effectiveness of the smaller incision, new generation (SING), implantable miniature telescope (IMT) in patients with moderate-severe central vision loss due to late-stage age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Following completion of informed consent, patients will be evaluated for eligibility to enroll into the study, including assessment of their best-corrected distance- and near- visual acuity with and without refraction, and also when using an external telescope simulator (ETS) to determine if they are likely to benefit from receiving the IMT. If eligible, they will be scheduled for out-patient surgery to implant the IMT during routine cataract surgery. Following implantation, patients will return for 5 post-operative follow-up visits over a period of approximately 12 months. Additionally, patients will have up to 12 rehabilitation/training visits with a low vision specialist

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 65 years of age at the Pre-operative Visit;
2. Have ETDRS BCDVA 0.9 to 1.6 logMAR (20/160 to 20/800) at the Pre-operative Visit caused by bilateral central scotomas associated with end-stage AMD;
3. Have bilateral retinal findings of geographic atrophy or disciform scar with foveal involvement, as determined by standard of care fluorescein angiography (FA) prior to the Pre-operative Visit;
4. Have been monitored by an eye care professional over the 6-month (or longer) period immediately prior to the Pre-operative Visit and have demonstrated no evidence of active choroidal neovascularization (CNV) prior to the Pre-operative Visit as demonstrated by the following:

   1. lack of need of treatment for CNV over the past 6 months, and
   2. lack of active exudative fluid on optical coherence tomography (OCT) over the past 6 months, and
   3. lack of Retinal hemorrhage on exam over a 6-month period or longer
5. Agree to participate in post-operative visual training

   For the Implanted Eye:
6. Have evidence of visually significant cataract at the Pre-operative Visit;
7. Agree to undergo pre-operative training and assessment (1 or more sessions) with low vision specialists (optometrist or occupational therapist) in the use of an external telescope model sufficient for patient assessment and patient must achieve at least a 5-letter ETDRS BCDVA improvement (0.1 logMAR) in the final assessment

   For the Non-Implanted Eye:
8. Have adequate peripheral vision at the Pre-operative Visit to allow navigation

Exclusion Criteria:

1. Have cognitive impairment that would interfere with the ability to understand and provide Informed Consent or prevent proper visual training/rehabilitation with the device;
2. Have any of the following conditions at the Pre-operative Visit:

   1. Stargardt macular dystrophy;
   2. Diabetic retinopathy;
   3. Untreated retinal tears;
   4. Retinal vascular disease;
   5. Optic nerve disease;
   6. History of retinal detachment;
   7. Intraocular tumor;
   8. Retinitis pigmentosa;
3. History of steroid-induced rise in intraocular pressure (IOP), uncontrolled glaucoma, or IOP >22 mmHg at the Pre-operative Visit;
4. Have known allergy to post-operative medications;
5. History of eye rubbing or an ocular condition that predisposes subject to eye rubbing;
6. Have had prior or expected ophthalmic surgery within 30 days of the Operative Visit;
7. Have any circumstance that, based on the Investigator's judgment, poses a concern for the subject's safety;
8. Any systemic disease or clinical evidence of any condition at the Pre-operative Visit which would make the subject in the opinion of the investigator unsuitable for the study;
9. Concurrent participation or prior participation in any investigative drug or device study within last 30 days prior to Pre-operative Visit

   For the Implanted Eye:
10. Have central anterior chamber depth (ACD) <3.0 mm from the posterior surface of the cornea (endothelium) to the anterior surface of the crystalline lens at the Pre-operative Visit;
11. Have an Endothelial Cell Density (ECD) below:

    1. 2,000 cells per millimeter, if 65-84 years old;
    2. 1,800 cells per millimeter, if 85 years old or greater (based on the lowest value of the three cell counts performed by technician at investigative site at the Pre-operative Visit)
12. Have a history of corneal stromal or endothelial dystrophies, including guttata;
13. Have Myopia > 6.0 D or Hyperopia > 4.0 D by Manifest Refraction at the Pre-operative Visit;
14. Have an Axial Length (AL) < 21 mm at the Pre-operative Visit;
15. Have a narrow angle defined as < grade 2 on the Schaffer scale at the Pre-operative Visit;
16. Ongoing Inflammatory ocular disease at the Pre-operative Visit;
17. Zonular weakness/instability of crystalline lens, or pseudoexfoliation at the Pre-operative Visit;
18. Have any condition at the Pre-operative Visit which in the judgement of the Investigator indicates that the haptics cannot be placed within the capsular bag during surgery;
19. Have had previous intraocular or corneal surgery, including any type of surgery for refractive or therapeutic purposes;

    For the Non-Implanted Eye:
20. Have ophthalmic pathology at the Pre-operative Visit that compromises the patient's peripheral vision based on the Investigator's judgment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Outcome | Approximately 12-months post-operatively (330-420 days)
  Proportion of study eyes with an improvement of 10 or more ETDRS letters (0.2 logMAR) in either BCDVA or BCNVA at Visit 5 (330 to 420 days post-operatively) compared to Pre-operative Visit
Primary Safety Outcome | Approximately 12-months post-operatively (330-420 days)
  Percent change in endothelial cell density (ECD) from Pre-operative Visit in study eyes at Visit 5 (330 to 420 days post-operatively)

SECONDARY OUTCOMES:
Best-corrected distance visual acuity (BCDVA) | Approximately 12-months post-operatively (330-420 days)
  Post-operative BCDVA in study eyes at Visit 5 (330 to 420 days post-operatively) compared to Pre-operative Visit
Best-corrected near visual acuity (BCNVA) | Approximately 12-months post-operatively (330-420 days)
  Post-operative BCNVA in study eyes at Visit 5 (330 to 420 days post-operatively) compared to Pre-operative Visit
Anterior Chamber Depth | Approximately 12-months post-operatively (330-420 days)
  Anterior Chamber Depth in study eyes, defined as the distance between the corneal endothelium and the front surface of the IMT, at Visit 5 (330 to 420 days post-operatively)
IMT position | Approximately 12-months post-operatively (330-420 days)
  IMT tilt and centration in study eyes at Visit 5 (330 to 420 days post-operatively)
Adverse Events | Approximately 12-months post-operatively (330-420 days)
  Rates of adverse events from Operative Visit through Visit 5 (330 to 420 days post-operatively)
Posterior Capsule Opacification | Approximately 12-months post-operatively (330-420 days)
  Rates of posterior capsule opacification in study eyes at post-operative visit 5 (330 to 420 days post-operatively)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Kammer, OD, PhD, Study Director — Samsara Vision Inc.
Locations (10):
- United States (10):
  - Loma Linda University, Loma Linda, California
  - Eye Physicians of Long Beach, Long Beach, California
  - Sarasota Retina Institute, Sarasota, Florida
  - Tallman Eye Associates, Lawrence, Massachusetts
  - Oakland Ophthalmic Surgery, Birmingham, Michigan
  - Vance Thompson Vision, Omaha, Nebraska
  - Atlantic Eye Physicians, Eatontown, New Jersey
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Cleveland Clinic | Cole Eye Institute, Cleveland, Ohio
  - Methodist Eye Associates | Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No